CLINICAL TRIAL: NCT00523718
Title: A Double-blind Study of Riluzole Augmentation in Serotonin Reuptake Inhibitor-refractory Obsessive-compulsive Disorder and Depression
Brief Title: Riluzole Augmentation in Treatment-refractory Obsessive-compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0509000614; R34MH083115 (NIH)
Record Dates: First submitted 2007-08-29; First posted 2007-08-31 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2020-03-06 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-compulsive Disorder; Ocd
Keywords: obsessive-compulsive disorder; OCD; glutamate; riluzole; augmentation; treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Compulsive Personality Disorder | interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- riluzole (Experimental): Patients randomized to this arm will receive riluzole augmentation, at a standard, fixed dose (50 mg bid), in addition to the medication regimen they are on at enrollment
  Interventions: Drug: riluzole
- placebo (Placebo Comparator): Patients randomized to this arm will receive placebo, formulated to be indistinguishable from riluzole, in addition to the medication regimen they are on at study enrollment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: riluzole — 50 mg PO bid, 12 weeks
  Other Names: Rilutek (Sanofi-Aventis)
  Arms: riluzole
Drug: placebo — placebo, 1 capsule PO bid, 12 weeks
  Arms: placebo

SUMMARY:
Obsessive-compulsive disorder (OCD) affects 2-3% of the population and leads to a great deal of suffering. Many patients benefit from established treatments, the mainstay of which are cognitive behavioral therapy and a group of antidepressant medications known as serotonin reuptake inhibitors. However, 20-30% of patients get minimal benefit from these established therapeutic strategies. New avenues of treatment are urgently needed.

Existing medications for obsessive-compulsive disorder affect the neurotransmitters serotonin or dopamine; but increasing evidence suggests that functional disruptions of a different neurotransmitter, glutamate, may contribute to some cases of OCD. The investigators are therefore interested in using medications that target glutamate as novel treatment options for those OCD patients who do not benefit from established treatments.

One such medication is the drug riluzole, which is FDA approved for amyotrophic lateral sclerosis (ALS), or Lou Gehrig's disease, but may be of benefit to patients with psychiatric disorders due to its ability to moderate excessive glutamate. In preliminary studies, in which the investigators treated patients with riluzole (in addition to their established pharmacological regimen) in an open-label fashion (that is, without a placebo-treated control group), the investigators have found about 40-50% of patients to substantially improve over 2-3 months.

While immensely promising, these preliminary studies do not prove riluzole is truly a new beneficial medication for the treatment of OCD; a more rigorous placebo-controlled trial is needed for that purpose. The investigators are therefore now recruiting patients to participate in a double-blind, placebo-controlled trial of riluzole, added to whatever other OCD medications they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) diagnosis of OCD, confirmed by Structured Clinical Interview for DSM-IV (SCID-IV); symptoms of at least 1 year duration
* moderate to severe OCD symptoms as measured by a score on the Yale-Brown Obsessive-Compulsive Scale (Y-BOCS) of 16 or greater
* documented failure of an adequate trial of a selective serotonin reuptake inhibitor (SSRI)
* agreement to engage in a reliable form of birth control (women only)

Exclusion Criteria:

* primary diagnosis of a psychotic disorder
* active substance abuse or dependence
* unstable medical condition
* prior exposure to riluzole
* prior psychosurgery
* pregnancy, breastfeeding, or intent to become pregnant during study
* liver function tests (LFTs) elevated to more than 2x the upper limit of normal
* evidence of active liver disease
* seizure disorder
* active suicidal ideation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Pittenger, MD, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale OCD Research Clinic, New Haven, Connecticut, United States

REFERENCES:
- [Background] Pittenger C, Krystal JH, Coric V. Glutamate-modulating drugs as novel pharmacotherapeutic agents in the treatment of obsessive-compulsive disorder. NeuroRx. 2006 Jan;3(1):69-81. doi: 10.1016/j.nurx.2005.12.006. PMID 16490414
- [Background] Coric V, Taskiran S, Pittenger C, Wasylink S, Mathalon DH, Valentine G, Saksa J, Wu YT, Gueorguieva R, Sanacora G, Malison RT, Krystal JH. Riluzole augmentation in treatment-resistant obsessive-compulsive disorder: an open-label trial. Biol Psychiatry. 2005 Sep 1;58(5):424-8. doi: 10.1016/j.biopsych.2005.04.043. PMID 15993857
- [Background] Pittenger C, Bloch MH, Williams K. Glutamate abnormalities in obsessive compulsive disorder: neurobiology, pathophysiology, and treatment. Pharmacol Ther. 2011 Dec;132(3):314-32. doi: 10.1016/j.pharmthera.2011.09.006. Epub 2011 Sep 22. PMID 21963369
- [Derived] Pittenger C, Bloch MH, Wasylink S, Billingslea E, Simpson R, Jakubovski E, Kelmendi B, Sanacora G, Coric V. Riluzole augmentation in treatment-refractory obsessive-compulsive disorder: a pilot randomized placebo-controlled trial. J Clin Psychiatry. 2015 Aug;76(8):1075-84. doi: 10.4088/JCP.14m09123. PMID 26214725
- See also: Yale OCD Research Clinic website — http://www.ocd.yale.edu
- See also: new Yale OCD Research Clinic website — http://psychiatry.yale.edu/ocd/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with selective serotonin reuptake inhibitor(SSRI)-refractory OCD were recruited through the Yale OCD Research Clinic between November 2006 and December 2012 using print and internet advertisements, community outreach, and physician referrals.
Pre-assignment Details: Forty subjects with treatment-refractory OCD were consented; 1 dropped out after consent, and one was excluded after it was revealed they were not taking an SSRI. These individuals were not randomized.
Period: Overall Study
Arm/Group | Riluzole | Placebo
Started | 20 | 18
Completed | 17 | 18
Not Completed | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Protocol Violation | 2 | 0

BASELINE CHARACTERISTICS:
Population: One individual was excluded from analysis (they were in the riluzole group) before unblinding due to a protocol violation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Riluzole | Placebo | Total
Number analyzed (Participants) | 19 | 18 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (3.2) | 36.4 (3.1) | 38.52 (13.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 9 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 19 | 16 | 35
  African American | 0 | 2 | 2
Y-BOCS baseline score [Mean (Standard Deviation); unit: units on a scale] — The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a test to rate the severity of obsessive-compulsive disorder (OCD) symptoms. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The results can be interpreted based on the total score:
  0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme.
  units on a scale | 30 (5.12) | 30.73 (5.81) | 30.37 (5.41)
HDRS baseline score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Depression Rating Scale (HDRS; also known as the HAM-D) is the most widely used clinician-administered depression assessment scale. The HAM-D 17-item scale ranges from 0 (normal) to >23 (very severe depression), with a maximum score of 52. The 24-item scale has a maximum score of 75. Severity of depression (e.g. "normal" or "very severe") is based upon the score in the first 17-items.
  units on a scale | 12.68 (6.89) | 13.05 (6.19) | 12.87 (6.46)
HARS baseline score [Mean (Standard Deviation); unit: units on a scale] — The Hamilton Anxiety Rating Scale (HARS or HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. Total score ranges from 0 to 56. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. A score of 25 to 30 indicates a moderate to severe anxiety severity. A score of 31 or greater represents very severe anxiety severity.
  units on a scale | 16.2 (7.35) | 15.95 (6.433) | 16.08 (6.80)

OUTCOME MEASURES:

1. Primary Outcome: Partial Responders by Yale-Brown Obsessive-Compulsive Scale (Y-BOCS)
Description: The Yale-Brown Obsessive Compulsive Scale (Y-BOCS) is a test to rate the severity of obsessive-compulsive disorder (OCD) symptoms. The scale is a clinician-rated, 10-item scale, each item rated from 0 (no symptoms) to 4 (extreme symptoms), yielding a total possible score range from 0 to 40. The results can be interpreted based on the total score:
  0-7 is sub-clinical; 8-15 is mild; 16-23 is moderate; 24-31 is severe; 32-40 is extreme.
  Improvement was defined apriori as a 25% improvement from baseline
Time Frame: 14 weeks
Measure: Number; unit: participants
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 18
participants | 5 | 2
Statistical Analysis 1: Comparison: Riluzole vs Placebo; Test type: Superiority or Other; p = .24, Chi-squared

2. Secondary Outcome: Average Hamilton Depression Inventory (HAM-D)
Description: The HDRS (also known as the HAM-D) is the most widely used clinician-administered depression assessment scale. The HAM-D 17-item scale ranges from 0 (normal) to >23 (very severe depression), with a maximum score of 52. The 24-item scale has a maximum score of 75. Severity of depression (e.g. "normal" or "very severe") is based upon the score in the first 17-items.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 11.941 (6.91) | 12.53 (5.67)

3. Secondary Outcome: Average Hamilton Anxiety Inventory (HAM-A)
Description: The Hamilton Anxiety Rating Scale (HARS or HAM-A) is a psychological questionnaire used by clinicians to rate the severity of a patient's anxiety. Total score ranges from 0 to 56. A score of 17 or less indicates mild anxiety severity. A score from 18 to 24 indicates mild to moderate anxiety severity. A score of 25 to 30 indicates a moderate to severe anxiety severity. A score of 31 or greater represents very severe anxiety severity.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 14.176 (6.80) | 14.263 (6.19)

4. Secondary Outcome: Clinical Global Impression (CGI) - Severity of Illness Item
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Considering total clinical experience, a patient is assessed on severity of mental illness at the time of rating 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Riluzole | Placebo
Number analyzed (Participants) | 19 | 18
units on a scale | 3.94 (1.09) | 3.95 (1.026)

ADVERSE EVENTS:
Description: Physical side effects were assessed by the Physical Symptom Checklist. Data from the Physical Symptom Checklist were not available for the first 4 patients randomized; the n for this analysis is therefore 16 for riluzole and 17 for placebo.
Arm/Group | Riluzole | Placebo
Serious Adverse Events (participants affected / at risk) | 1/19 | 1/18
Other Adverse Events (participants affected / at risk) | 7/16 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riluzole (N=19) | Placebo (N=18)
Passively Suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Overdose of Narcotics (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Riluzole (N=16) | Placebo (N=17)
Nausea (Gastrointestinal disorders) | 3 | 1
Poor Coordination (Nervous system disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 1 | 6
Pounding Heart Beat (Cardiac disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes